CLINICAL TRIAL: NCT00033605
Title: Phase III Double-Blind Study Of Depot Octreotide Versus Placebo In The Prevention Of Acute Diarrhea In Patients Receiving Pelvic Radiation Therapy
Brief Title: Octreotide in Preventing Diarrhea in Patients Who Are Undergoing Radiation Therapy to the Pelvis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N00CA; CDR0000069304 (Registry Identifier: PDQ (Physician Data Query)); NCI-P02-0221
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Cervical Cancer; Colorectal Cancer; Diarrhea; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Prostate Cancer; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific; Vaginal Cancer; Vulvar Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Colorectal Neoplasms; Diarrhea; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Sarcoma; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Octreotide; Radiation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- octreotide + radiation (Experimental): Patients receive short-acting octreotide subcutaneously (SC) on day 1 and long-acting octreotide intramuscularly (IM) on days 2 and 29.
  Treatment continues in the absence of unacceptable toxicity or the development of severe diarrhea.
  Patients complete a bowel function questionnaire at baseline, weekly during radiotherapy, and then weekly for 4 weeks and at 1 and 2 years after completion of radiotherapy.
  Patients are followed weekly for 4 weeks and then at 1 and 2 years.
  Interventions: Drug: octreotide acetate; Radiation: radiation
- placebo + radiation (Active Comparator): Patients receive placebo SC on day 1 and IM on days 2 and 29. Treatment continues in the absence of unacceptable toxicity or the development of severe diarrhea.
  Patients complete a bowel function questionnaire at baseline, weekly during radiotherapy, and then weekly for 4 weeks and at 1 and 2 years after completion of radiotherapy.
  Patients are followed weekly for 4 weeks and then at 1 and 2 years.
  Interventions: Other: placebo; Radiation: radiation

INTERVENTIONS:
Drug: octreotide acetate
  Arms: octreotide + radiation
Other: placebo
  Arms: placebo + radiation
Radiation: radiation

SUMMARY:
RATIONALE: Octreotide may be effective in preventing or controlling diarrhea in patients who are undergoing radiation therapy to the pelvis. It is not yet known whether octreotide is effective for diarrhea.

PURPOSE: Randomized phase III trial to determine the effectiveness of octreotide in preventing diarrhea in patients who are undergoing radiation therapy to the pelvis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of octreotide in reducing acute treatment-related diarrhea in patients receiving external-beam radiotherapy to the pelvis.
* Determine the effectiveness of this drug in reducing chronic treatment-related bowel dysfunction in these patients.
* Determine the toxicity of this drug in these patients.
* Assess the importance that these patients attach to various measures of bowel function.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to prior anterior resection of the rectum (yes vs no), total planned cumulative dose of radiotherapy, including boost fields (4,500-5,350 cGy vs 5,351-6,000 cGy vs more than 6,000 cGy), use of concurrent fluorouracil (none vs bolus vs continuous infusion), use of concurrent leucovorin calcium (yes vs no), use of concurrent cisplatin (yes vs no), superior border of initial field (at or inferior to the L4-5 interspace vs superior to the L4-5 interspace), planned intracavitary brachytherapy (yes vs no), and primary site of disease (rectal cancer vs prostate cancer vs gynecological cancer vs other). Beginning no later than the fourth day of radiotherapy, patients are randomized to one of two treatment arms.

* Arm I: Patients receive short-acting octreotide subcutaneously (SC) on day 1 and long-acting octreotide intramuscularly (IM) on days 2 and 29.
* Arm II: Patients receive placebo SC on day 1 and IM on days 2 and 29. In both arms, treatment continues in the absence of unacceptable toxicity or the development of severe diarrhea.

Patients complete a bowel function questionnaire at baseline, weekly during radiotherapy, and then weekly for 4 weeks and at 1 and 2 years after completion of radiotherapy.

Patients are followed weekly for 4 weeks and then at 1 and 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer in the pelvis
* Plan to receive continuous definitive or adjuvant external-beam radiotherapy to the pelvis or pelvis and para-aortic lymph nodes (total planned dose of 4,500-5,350 cGy)

  * Entire pelvis must be encompassed by planned radiotherapy field (superior border not inferior to the most inferior aspect of sacroiliac joints)
  * Portions of rectum may have special blocking depending on disease site
  * Planned treatment for once-daily radiotherapy 4-5 times a week (planned daily dose 170-210 cGy)
  * No planned split-course radiotherapy
  * No planned interstitial brachytherapy prior to completion of external-beam radiotherapy
  * Planned intracavitary radiotherapy allowed
  * No planned cytotoxic chemotherapy agents concurrently with radiotherapy except fluorouracil with or without leucovorin calcium or cisplatin
  * Entered on study before the third radiotherapy fraction
* No current or prior metastases beyond pelvic or para-aortic lymph nodes
* No grade 3 or greater diarrhea, rectal bleeding, or abdominal cramping prior to radiotherapy
* No incontinence of stool

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Renal:

* No chronic renal failure
* Creatinine less than 2 times upper limit of normal (for patients with history of renal disease)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known allergy to octreotide
* No history of inflammatory bowel disease
* No other concurrent medical condition that would preclude study participation
* No history of cholecystitis unless prior cholecystectomy

PRIOR CONCURRENT THERAPY:

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to the pelvis

Surgery:

* See Disease Characteristics
* No prior abdominal-perineal resection, Hartmann procedure, or other surgical procedure resulting in non-functioning rectum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2002-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Reduction of diarrhea as measured by NCI CTC version 2.0 weekly during pelvic radiotherapy | Up to 2 years

SECONDARY OUTCOMES:
Reduction of patient-reported bowel dysfunction as assessed by the bowel function questionnaire weekly during radiotherapy, weekly for 4 weeks after radiotherapy, and 12 and 24 months after completion of radiotherapy | Up to 2 years
Toxicity as assessed by NCI CTC version 2.0 weekly during pelvic radiotherapy | Up to 2 years
Importance that patients attach to various measures of bowel dysfunction as assessed by questionnaire at week 4 of radiotherapy and at 12 and 24 months after completion of radiotherapy | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James A. Martenson, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Martenson JA, Halyard MY, Sloan JA, Proulx GM, Miller RC, Deming RL, Dick SJ, Johnson HA, Tai TH, Zhu AW, Keit J, Stien KJ, Atherton PJ. Phase III, double-blind study of depot octreotide versus placebo in the prevention of acute diarrhea in patients receiving pelvic radiation therapy: results of North Central Cancer Treatment Group N00CA. J Clin Oncol. 2008 Nov 10;26(32):5248-53. doi: 10.1200/JCO.2008.17.1546. Epub 2008 Sep 2. PMID 18768432